CLINICAL TRIAL: NCT03373383
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose Finding Study to Evaluate the Efficacy and Safety of Padsevonil as Adjunctive Treatment of Focal-Onset Seizures in Adult Subjects With Drug-Resistant Epilepsy
Brief Title: Study to Test the Efficacy and Safety of Padsevonil as Adjunctive Treatment of Focal-onset Seizures in Adults With Drug-resistant Epilepsy
Acronym: ARISE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EP0091; 2017-003200-48 (EudraCT Number)
Record Dates: First submitted 2017-12-07; First posted 2017-12-14 (Actual); Results first posted 2021-04-09 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Drug-resistant Epilepsy; Focal-Onset Seizures
Keywords: Epilepsy; Padsevonil
MeSH Terms: conditions — Drug Resistant Epilepsy; Seizures; Epilepsy | interventions — padsevonil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Padsevonil dosing regimen 1 (Experimental): Subjects will be randomized to receive a combination of tablets of Padsevonil and Placebo (as appropriate) to maintain the blinding.
  Interventions: Drug: Padsevonil; Other: Placebo
- Padsevonil dosing regimen 2 (Experimental): Subjects will be randomized to receive a combination of tablets of Padsevonil and Placebo (as appropriate) to maintain the blinding.
  Interventions: Drug: Padsevonil; Other: Placebo
- Padsevonil dosing regimen 3 (Experimental): Subjects will be randomized to receive a combination of tablets of Padsevonil and Placebo (as appropriate) to maintain the blinding.
  Interventions: Drug: Padsevonil; Other: Placebo
- Padsevonil dosing regimen 4 (Experimental): Subjects will be randomized to receive a combination of tablets of Padsevonil and Placebo (as appropriate) to maintain the blinding.
  Interventions: Drug: Padsevonil; Other: Placebo
- Placebo (Placebo Comparator): Subjects randomized to the placebo group will receive a combination of several Placebo tablets to maintain the blinding.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Padsevonil — Padsevonil in different dosages.
  Arms: Padsevonil dosing regimen 1; Padsevonil dosing regimen 2; Padsevonil dosing regimen 3; Padsevonil dosing regimen 4
Other: Placebo — Placebo will be provided matching Padsevonil.

SUMMARY:
The purpose of the study is to characterize the dose-response relationship with respect to efficacy of Padsevonil administered concomitantly with up to 3 anti-epileptic drugs (AEDs) for treatment of observable focal-onset seizures in subjects with drug-resistant epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of focal epilepsy per 1989 International League Against Epilepsy (ILAE) criteria at least 3 years before study entry
* Subject has failed to achieve seizure control with 4 tolerated and appropriately chosen prior antiepileptic drugs (AED), including past and ongoing treatment, that were individually optimized for adequate dose and duration. Prior discontinued AED treatment would need to be assessed by the Investigator considering the patient medical records and patient and/or caregiver interview. 'Prior AED' is defined as all past and ongoing AED treatments with a start date before the Screening Visit (Visit 1)
* Average of >= 4 spontaneous and observable focal seizures (type IA1 (i.e. focal aware), IB (i.e. focal impaired awareness), IC (i.e. focal to bilateral tonic-clonic)) per month
* Current treatment with an individually optimized and stable dose of at least 1 and up to 3 AEDs for the 8 weeks prior to the Screening Visit with or without additional Vagus Nerve Stimulation (VNS) or other neurostimulation treatments

Exclusion Criteria:

* Subject has a history of or signs of generalized or combined generalized and focal epilepsy
* Cluster seizures which are uncountable in the previous 8 weeks before study entry and during 4 weeks prospective baseline
* Current treatment with carbamazepine, phenytoin, primidone, phenobarbital
* Current treatment/ use of (non-AED) prescription, nonprescription, dietary (eg, grapefruit or passion fruit), or herbal products that are potent inducers or inhibitors of the CYP3A4 or 2C19 pathway for 2 weeks (or 5 half-lives, whichever is longer) prior to the Baseline Visit
* Subjects taking sensitive substrates of CYP2C19 for 2 weeks (or 5 half-lives, whichever is longer) prior to the Baseline Visit
* Subject has been taking vigabatrin less than 2 years at study entry
* Subject has been taking felbamate for less than 12 months
* Subject taking retigabine for less than 4 years
* Current treatment with benzodiazepines (i.e. GABA-A-ergic drugs like zolpidem, zaleplon, or zopiclone, excluding GABA-A-ergic AEDs) <3 times per week for emergencies
* Subject has a current medical condition that occurred within the last 12 months which, in the opinion of the investigator, could compromise his/her safety or ability to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 411 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (148):
- United States (27):
  - Ep0091 839, Chandler, Arizona
  - Ep0091 810, Little Rock, Arkansas
  - Ep0091 815, La Jolla, California
  - Ep0091 801, San Francisco, California
  - Ep0091 845, Washington D.C., District of Columbia
  - Ep0091 809, Ocala, Florida
  - Ep0091 823, Orlando, Florida
  - Ep0091 825, Port Charlotte, Florida
  - Ep0091 820, Tallahassee, Florida
  - Ep0091 873, Atlanta, Georgia
  - Ep0091 803, Honolulu, Hawaii
  - Ep0091 832, Peoria, Illinois
  - Ep0091 822, Baltimore, Maryland
  - Ep0091 818, Bethesda, Maryland
  - Ep0091 817, Saint Paul, Minnesota
  - Ep0091 806, Hackensack, New Jersey
  - Ep0091 827, New York, New York
  - Ep0091 800, Philadelphia, Pennsylvania
  - Ep0091 802, Philadelphia, Pennsylvania
  - Ep0091 838, Cordova, Tennessee
  - Ep0091 835, Nashville, Tennessee
  - Ep0091 805, Austin, Texas
  - Ep0091 844, Austin, Texas
  - Ep0091 836, Dallas, Texas
  - Ep0091 830, Dallas, Texas
  - Ep0091 824, Round Rock, Texas
  - Ep0091 870, San Antonio, Texas
- Australia (8):
  - Ep0091 855, Box Hill
  - Ep0091 857, Clayton
  - Ep0091 850, Fitzroy
  - Ep0091 859, Herston
  - Ep0091 852, Melbourne
  - Ep0091 853, Melbourne
  - Ep0091 856, Randwick
  - Ep0091 854, Westmead
- Belgium (4):
  - Ep0091 102, Bruges
  - Ep0091 101, Brussels
  - Ep0091 105, Ghent
  - Ep0091 100, Leuven
- Bulgaria (6):
  - Ep0091 150, Blagoevgrad
  - Ep0091 151, Pleven
  - Ep0091 153, Pleven
  - Ep0091 152, Sofia
  - Ep0091 154, Sofia
  - Ep0091 155, Sofia
- Canada (3):
  - Ep0091 200, Greenfield Park
  - Ep0091 205, London
  - Ep0091 201, Montreal
- Czechia (6):
  - Ep0091 254, Brno
  - Ep0091 255, Ostrava-Poruba
  - Ep0091 250, Prague
  - Ep0091 251, Prague
  - Ep0091 252, Prague
  - Ep0091 253, Prague
- France (7):
  - Ep0091 307, Clermont-Ferrand
  - Ep0091 309, Dijon
  - Ep0091 300, Lille
  - Ep0091 302, Montpellier
  - Ep0091 305, Paris
  - Ep0091 303, Rennes
  - Ep0091 306, Toulouse
- Germany (18):
  - Ep0091 361, Bad Neustadt an der Saale
  - Ep0091 365, Berlin
  - Ep0091 362, Bernau
  - Ep0091 363, Bielefeld
  - Ep0091 358, Bonn
  - Ep0091 350, Frankfurt am Main
  - Ep0091 360, Freiburg im Breisgau
  - Ep0091 364, Hamburg
  - Ep0091 368, Jena
  - Ep0091 366, Kork
  - Ep0091 357, Leipzig
  - Ep0091 353, Marburg
  - Ep0091 354, München
  - Ep0091 351, Münster
  - Ep0091 356, Osnabrück
  - Ep0091 367, Ravensburg
  - Ep0091 301, Strausberg
  - Ep0091 352, Tübingen
- Hungary (3):
  - Ep0091 400, Budapest
  - Ep0091 403, Budapest
  - Ep0091 402, Debrecen
- Italy (11):
  - Ep0091 462, Bologna
  - Ep0091 450, Cagliari
  - Ep0091 461, Foggia
  - Ep0091 452, Milan
  - Ep0091 459, Pavia
  - Ep0091 453, Perugia
  - Ep0091 458, Pozzilli
  - Ep0091 454, Reggio Calabria
  - Ep0091 455, Roma
  - Ep0091 457, Roma
  - Ep0091 460, Roma
- Japan (11):
  - Ep0091 501, Asaka
  - Ep0091 511, Fukuoka
  - Ep0091 505, Hiroshima
  - Ep0091 513, Hōfu
  - Ep0091 507, Itami
  - Ep0091 503, Kodaira
  - Ep0091 514, Kyoto
  - Ep0091 512, Nagakute
  - Ep0091 510, Niigata
  - Ep0091 515, Saitama
  - Ep0091 509, Shizuoka
- Lithuania (3):
  - Ep0091 703, Kaunas
  - Ep0091 701, Vilnius
  - Ep0091 702, Vilnius
- Mexico (2):
  - Ep0091 553, Culiacán
  - Ep0091 552, Mexico City
- Poland (10):
  - Ep0091 601, Gdansk
  - Ep0091 607, Grodzisk Mazowiecki
  - Ep0091 605, Katowice
  - Ep0091 608, Katowice
  - Ep0091 603, Krakow
  - Ep0091 604, Lublin
  - Ep0091 606, Nowa Sól
  - Ep0091 600, Poznan
  - Ep0091 609, Poznan
  - Ep0091 602, Świdnik
- Ep0091 952, Santa Maria da Feira, Portugal
- Slovakia (2):
  - Ep0091 004, Bardejov
  - Ep0091 001, Hlohovec
- Spain (17):
  - Ep0091 662, Alicante
  - Ep0091 651, Barcelona
  - Ep0091 652, Barcelona
  - Ep0091 658, Barcelona
  - Ep0091 664, Barcelona
  - Ep0091 668, Bilbao
  - Ep0091 666, Córdoba
  - Ep0091 650, Madrid
  - Ep0091 656, Madrid
  - Ep0091 660, Madrid
  - Ep0091 661, Madrid
  - Ep0091 659, Málaga
  - Ep0091 663, Seville
  - Ep0091 665, Terrassa
  - Ep0091 657, Valencia
  - Ep0091 667, Valencia
  - Ep0091 653, Valladolid
- Turkey (Türkiye) (3):
  - Ep0091 904, Eskişehir
  - Ep0091 900, Istanbul
  - Ep0091 901, Istanbul
- United Kingdom (6):
  - Ep0091 752, Birmingham
  - Ep0091 751, Cardiff
  - Ep0091 756, Inverness
  - Ep0091 757, London
  - Ep0091 750, Manchester
  - Ep0091 753, Swansea

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: http://www.Vivli.org

REFERENCES:
- [Result] Rademacher M, Toledo M, Van Paesschen W, Liow KK, Milanov IG, Esch ML, Wang N, MacPherson M, Byrnes WJ, Minh TDC, Webster E, Werhahn KJ. Efficacy and safety of adjunctive padsevonil in adults with drug-resistant focal epilepsy: Results from two double-blind, randomized, placebo-controlled trials. Epilepsia Open. 2022 Dec;7(4):758-770. doi: 10.1002/epi4.12656. Epub 2022 Oct 22. PMID 36176044
- [Result] Kramer H, Bicer C, Otoul C, Rospo C, Macpherson M, Watling M, Bani M, Sciberras D, Chanteux H. Clinical Bridging Studies and Modeling Approach for Implementation of a Patient Centric Sampling Technique in Padsevonil Clinical Development. AAPS J. 2023 Nov 16;26(1):1. doi: 10.1208/s12248-023-00866-7. PMID 37973662

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in February 2018 and concluded in January 2020.
Pre-assignment Details: The study included: a 4-week Baseline Period, a 16-week Treatment Period, a 4-week Taper Period (for participants who discontinued or choose not to enroll in the open-label extension study) and a Safety Follow-up Period. Participants continuing to the OLE study had a 3-week Conversion Period.
  Participant Flow refers to the Randomized Set.
Groups:
- Placebo: Participants randomized to the placebo group received 5-6 placebo tablets to maintain the blinding up to week 19.
- Padsevonil 50mg BID: Participants were randomized to receive a combination of tablets of padsevonil 50 milligrams (mg) and placebo (as appropriate) to maintain the blinding, twice daily (bid) up to week 19
- Padsevonil 100mg BID: Participants were randomized to receive a combination of tablets of padsevonil 100 mg and placebo (as appropriate) to maintain the blinding, bid up to week 19.
- Padsevonil 200mg BID: Participants were randomized to receive a combination of tablets of padsevonil 200 mg and placebo (as appropriate) to maintain the blinding, bid up to week 19.
- Padsevonil 400mg BID: Participants were randomized to receive a combination of tablets of padsevonil 400 mg and placebo (as appropriate) to maintain the blinding, bid up to week 19.
Period: Treatment Period: Wk0-16
Arm/Group | Placebo | Padsevonil 50mg BID | Padsevonil 100mg BID | Padsevonil 200mg BID | Padsevonil 400mg BID
Started | 83 | 81 | 83 | 82 | 82
Completed Titration and Stabilization | 78 | 72 | 71 | 68 | 65
Completed Maintenance Period | 70 | 66 | 68 | 61 | 58
Had Taper and Safety Follow-up | 6 | 11 | 8 | 18 | 21
Completed | 70 | 66 | 68 | 61 | 58
Not Completed | 13 | 15 | 15 | 21 | 24
Not completed — Adverse Event | 7 | 6 | 11 | 15 | 21
Not completed — Lack of Efficacy | 2 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 4 | 2 | 1 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 2 | 3 | 3
Not completed — As advised by the sponsor | 0 | 1 | 0 | 0 | 0
Not completed — By opinion of investigator | 0 | 0 | 0 | 1 | 0
Not completed — Sponsor decision | 0 | 0 | 0 | 1 | 0
Period: Post-Treatment Period: Wk16-23
Arm/Group | Placebo | Padsevonil 50mg BID | Padsevonil 100mg BID | Padsevonil 200mg BID | Padsevonil 400mg BID
Started | 70 | 66 | 68 | 61 | 58
Started Conversion Period | 69 | 64 | 66 | 55 | 57
Completed Conversion Period | 68 | 64 | 66 | 55 | 57
Had Taper and Safety Follow-up | 3 | 3 | 3 | 6 | 1
Enrolled in EP0093 | 67 | 63 | 65 | 55 | 57
Completed | 69 | 66 | 68 | 61 | 58
Not Completed | 1 | 0 | 0 | 0 | 0
Not completed — Participant decided not to roll over | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics refer to the Randomized Set (RS) consisting of all participants randomized into the study.
Arm/Group | Placebo | Padsevonil 50mg BID | Padsevonil 100mg BID | Padsevonil 200mg BID | Padsevonil 400mg BID | Total Title
Number analyzed (Participants) | 83 | 81 | 83 | 82 | 82 | 411
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 2 | 1 | 1 | 4
  Between 18 and 65 years | 82 | 76 | 80 | 79 | 80 | 397
  >=65 years | 1 | 5 | 1 | 2 | 1 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.0 (12.9) | 42.5 (11.6) | 36.9 (13.1) | 40.9 (12.0) | 38.8 (12.1) | 39.8 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 46 | 47 | 51 | 43 | 235
  Male | 35 | 35 | 36 | 31 | 39 | 176
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 1 | 2 | 0 | 5
  Asian | 7 | 7 | 5 | 7 | 7 | 33
  Black or African American | 2 | 1 | 1 | 2 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 1 | 1 | 1 | 5
  White | 69 | 69 | 73 | 69 | 71 | 351
  Other/mixed | 3 | 2 | 2 | 1 | 1 | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in Log-transformed Observable Focal Onset Seizure Frequency From Baseline Over the 12 Week Maintenance Period
Description: During the study, participants kept diaries to record daily seizure activity. Seizure frequency refers to 28-day adjusted frequency. Seizure frequency was based on investigator assessment of participants' reports of daily seizure type and frequency. Observable focal-onset seizures refer to Type IA1, IB, and IC (ILAE Classification of Epileptic Seizures, 1981). Based on ANCOVA on change in log-transformed, 28-day adjusted seizure frequency from Baseline with treatment group as the main factor, Baseline log-transformed seizure frequency as a continuous covariate, Baseline SV2A use (yes or no) and Region (Europe, Non-Europe) as categorical factors.
Time Frame: From Baseline over the 12 Week Maintenance Period
Population: The Full Analysis Set (FAS) consisted of all study participants in the RS who were administered at least 1 dose or a partial dose of IMP and had Baseline and at least 1 post-Baseline seizure frequency data during the 16-week Treatment Period.
Measure: Least Squares Mean (95% Confidence Interval); unit: loge seizures per 28 days
Groups:
- Placebo (FAS): Participants randomized to the placebo group received 5-6 placebo tablets to maintain the blinding up to week 19. Participants formed the Full Analysis Set (FAS).
- Padsevonil 50mg BID (FAS): Participants were randomized to receive a combination of tablets of padsevonil 50 mg and placebo (as appropriate) to maintain the blinding, bid up to week 19. Participants formed the FAS.
- Padsevonil 100mg BID (FAS): Participants were randomized to receive a combination of tablets of padsevonil 100 mg and placebo (as appropriate) to maintain the blinding, bid up to week 19. Participants formed the FAS.
- Padsevonil 200mg BID (FAS): Participants were randomized to receive a combination of tablets of padsevonil 200 mg and placebo (as appropriate) to maintain the blinding, bid up to week 19. Participants formed the FAS.
- Padsevonil 400mg BID (FAS): Participants were randomized to receive a combination of tablets of padsevonil 400 mg and placebo (as appropriate) to maintain the blinding, bid up to week 19. Participants formed the FAS.
Arm/Group | Placebo (FAS) | Padsevonil 50mg BID (FAS) | Padsevonil 100mg BID (FAS) | Padsevonil 200mg BID (FAS) | Padsevonil 400mg BID (FAS)
Number analyzed (Participants) | 81 | 80 | 82 | 81 | 81
loge seizures per 28 days | -0.27585 [-0.44311 to -0.10858] | -0.46424 [-0.63276 to -0.29573] | -0.48804 [-0.65436 to -0.32172] | -0.48960 [-0.65734 to -0.32187] | -0.40831 [-0.57485 to -0.24177]
Statistical Analysis 1: Comparison: Placebo (FAS) vs Padsevonil 50mg BID (FAS); Percent reduction over placebo was calculated as 100*(1-exp(diff)), where diff was the model estimate of the log ratio between each PSL group and placebo group; Test type: Superiority; p = 0.102, ANCOVA — Adjusted p-values were from the Hochberg step-up procedure within SAS® Proc Multtest to control Type I error; Percent reduction = 17.2, 95% CI 2-sided [-3.8 to 33.9]
Statistical Analysis 2: Comparison: Placebo (FAS) vs Padsevonil 100mg BID (FAS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.064, ANCOVA — Adjusted p-values were from the Hochberg step-up procedure within SAS® Proc Multtest to control Type I error; Percent reduction = 19.1, 95% CI 2-sided [-1.2 to 35.4]
Statistical Analysis 3: Comparison: Placebo (FAS) vs Padsevonil 200mg BID (FAS); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.063, ANCOVA — Adjusted p-values were from the Hochberg step-up procedure within SAS® Proc Multtest to control Type I error; Percent reduction = 19.2, 95% CI 2-sided [-1.2 to 35.5]
Statistical Analysis 4: Comparison: Placebo (FAS) vs Padsevonil 400mg BID (FAS); Percent reduction over placebo was calculated as 100*(1-exp[diff]), where diff was the model estimate of the log ratio between each PSL group and placebo group; Test type: Superiority; p = 0.248, ANCOVA — Adjusted p-values were from the Hochberg step-up procedure within SAS® Proc Multtest to control Type I error; Percent reduction = 12.4, 95% CI 2-sided [-9.7 to 30.1]

2. Secondary Outcome: 75 % Responder Rate Over the 12 Week Maintenance Period
Description: The 75% responder rate, where a responder is a participant experiencing a ≥75% reduction in observable focal-onset seizure frequency from Baseline, over the 12-Week Maintenance Period.
Time Frame: End of Maintenance Period (Week 16) following 3 Weeks of titration and 1 Week stabilization
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (FAS) | Padsevonil 50mg BID (FAS) | Padsevonil 100mg BID (FAS) | Padsevonil 200mg BID (FAS) | Padsevonil 400mg BID (FAS)
Number analyzed (Participants) | 81 | 80 | 82 | 81 | 81
percentage of participants | 6.2 | 13.8 | 12.2 | 11.1 | 16.0
Statistical Analysis 1: Comparison: Placebo (FAS) vs Padsevonil 50mg BID (FAS); PSL dose/Placebo was calculated using logistic regression with categorical factors for treatment group, Region (Europe, Non-Europe), Baseline SV2A use (0, 1) and log-transformed Baseline seizure frequency as a continuous covariate; Test type: Superiority; p = 0.081, Regression, Logistic — Nominal p-values were not adjusted for multiplicity; Odds Ratio (OR) = 2.72, 95% CI 2-sided [0.88 to 8.39]
Statistical Analysis 2: Comparison: Placebo (FAS) vs Padsevonil 100mg BID (FAS); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.137, Regression, Logistic — Nominal p-values were not adjusted for multiplicity; Odds Ratio (OR) = 2.37, 95% CI 2-sided [0.76 to 7.41]
Statistical Analysis 3: Comparison: Placebo (FAS) vs Padsevonil 200mg BID (FAS); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.192, Regression, Logistic — Nominal p-values were not adjusted for multiplicity; Odds Ratio (OR) = 2.16, 95% CI 2-sided [0.68 to 6.89]
Statistical Analysis 4: Comparison: Placebo (FAS) vs Padsevonil 400mg BID (FAS); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.041, Regression, Logistic — Nominal p-values were not adjusted for multiplicity; Odds Ratio (OR) = 3.14, 95% CI 2-sided [1.05 to 9.42]

3. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs) Reported by the Subject and/or Caregiver or Observed by the Investigator During the Entire Study
Description: An Adverse Event is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment.
Time Frame: From Baseline until Safety Follow-Up (up to Week 23)
Population: The Safety Set consisted of all study participants who were administered at least 1 dose or a partial dose of IMP.
Measure: Number; unit: percentage of participants
Groups:
- Placebo (SS): Participants randomized to the placebo group received 5-6 placebo tablets to maintain the blinding up to week 19. Participants formed the Safety Set (SS).
- Padsevonil 50mg BID (SS): Participants were randomized to receive a combination of tablets of padsevonil 50 mg and Placebo (as appropriate) to maintain the blinding, bid up to week 19. Participants formed the SS.
- Padsevonil 100mg BID (SS): Participants were randomized to receive a combination of tablets of padsevonil 100 mg and placebo (as appropriate) to maintain the blinding, bid up to week 19. Participants formed the SS.
- Padsevonil 200mg BID (SS): Participants were randomized to receive a combination of tablets of padsevonil 200 mg and placebo (as appropriate) to maintain the blinding, bid up to week 19. Participants formed the SS.
- Padsevonil 400mg BID (SS): Participants were randomized to receive tablets of padsevonil 400 mg and placebo (as appropriate) to maintain the blinding, bid up to week 19. Participants formed the SS.
Arm/Group | Placebo (SS) | Padsevonil 50mg BID (SS) | Padsevonil 100mg BID (SS) | Padsevonil 200mg BID (SS) | Padsevonil 400mg BID (SS)
Number analyzed (Participants) | 83 | 81 | 83 | 82 | 81
percentage of participants | 78.3 | 84.0 | 80.7 | 75.6 | 92.6

4. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs) Leading to Study Withdrawal
Description: as for outcome 3
Time Frame: From Baseline until Safety Follow-Up (up to Week 23)
Population: The Safety Set consisted of all study participants who were administered at least 1 dose or a partial dose of IMP.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (SS) | Padsevonil 50mg BID (SS) | Padsevonil 100mg BID (SS) | Padsevonil 200mg BID (SS) | Padsevonil 400mg BID (SS)
Number analyzed (Participants) | 83 | 81 | 83 | 82 | 81
percentage of participants | 8.4 | 7.4 | 12.0 | 18.3 | 25.9

5. Primary Outcome: Percentage of Participants With Treatment-Emergent Serious Adverse Events (SAEs) During the Entire Study
Description: A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose:
  * Results in death
  * Is life-threatening
  * Requires in patient hospitalization or prolongation of existing hospitalization
  * Is a congenital anomaly or birth defect
  * Is an infection that requires treatment parenteral antibiotics
  * Other important medical events which based on medical or scientific judgement may jeopardize the patients, or may require medical or surgical intervention to prevent any of the above.
Time Frame: From Baseline until Safety Follow-Up (up to Week 23)
Population: The Safety Set consisted of all study participants who were administered at least 1 dose or a partial dose of IMP.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (SS) | Padsevonil 50mg BID (SS) | Padsevonil 100mg BID (SS) | Padsevonil 200mg BID (SS) | Padsevonil 400mg BID (SS)
Number analyzed (Participants) | 83 | 81 | 83 | 82 | 81
percentage of participants | 4.8 | 7.4 | 4.8 | 6.1 | 6.2

6. Secondary Outcome: 50 % Responder Rate Over the 12 Week Maintenance Period
Description: The 50% responder rate, where a responder was a participant experiencing a ≥50% reduction in observable focal-onset seizure frequency from Baseline, over the 12-Week Maintenance Period.
Time Frame: End of Maintenance Period (Week 16) following 3 Weeks of titration and 1 Week stabilization
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (FAS) | Padsevonil 50mg BID (FAS) | Padsevonil 100mg BID (FAS) | Padsevonil 200mg BID (FAS) | Padsevonil 400mg BID (FAS)
Number analyzed (Participants) | 81 | 80 | 82 | 81 | 81
percentage of participants | 21.0 | 33.8 | 31.7 | 25.9 | 32.1
Statistical Analysis 1: Comparison: Placebo (FAS) vs Padsevonil 50mg BID (FAS); PSL dose/placebo calculated using logistic regression with categorical factors for treatment group (each PSL dose group referenced to the placebo group), region (Europe, Non-Europe), Baseline SV2A use (0, 1) and log-transformed Baseline seizure frequency as a continuous covariate; Test type: Superiority; p = 0.045, Regression, Logistic — Nominal p-values were not adjusted for multiplicity; Odds Ratio (OR) = 2.09, 95% CI 2-sided [1.02 to 4.30]
Statistical Analysis 2: Comparison: Placebo (FAS) vs Padsevonil 100mg BID (FAS); [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.079, Regression, Logistic — Nominal p-values were not adjusted for multiplicity; Odds Ratio (OR) = 1.91, 95% CI 2-sided [0.93 to 3.93]
Statistical Analysis 3: Comparison: Placebo (FAS) vs Padsevonil 200mg BID (FAS); [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.338, Regression, Logistic — Nominal p-values were not adjusted for multiplicity; Odds Ratio (OR) = 1.44, 95% CI 2-sided [0.68 to 3.02]
Statistical Analysis 4: Comparison: Placebo (FAS) vs Padsevonil 400mg BID (FAS); PSL dose/Placebo calculated using logistic regression with categorical factors for treatment group, Region (Europe, Non-Europe), Baseline SV2A use (0, 1) and log-transformed Baseline seizure frequency as a continuous covariate; Test type: Superiority; p = 0.087, Regression, Logistic — Nominal p-values were not adjusted for multiplicity; Odds Ratio (OR) = 1.88, 95% CI 2-sided [0.91 to 3.87]

7. Secondary Outcome: Percent Change in Observable Focal-onset Seizure Frequency From Baseline Over the 12 Week Maintenance Period
Description: During the study, participants kept diaries to record daily seizure activity. The percentage of participants who experienced a 50 % or greater reduction in seizure frequency per 28 days relative to Baseline (responders) was assessed.
Time Frame: End of Maintenance Period (Week 16) following 3 Weeks of titration and 1 Week stabilization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo (FAS) | Padsevonil 50mg BID (FAS) | Padsevonil 100mg BID (FAS) | Padsevonil 200mg BID (FAS) | Padsevonil 400mg BID (FAS)
Number analyzed (Participants) | 81 | 80 | 82 | 81 | 81
percent change | 12.49 (58.26) | 24.70 (46.62) | 25.25 (51.73) | 20.79 (66.54) | 15.79 (67.55)
Statistical Analysis 1: Comparison: Placebo (FAS) vs Padsevonil 50mg BID (FAS); Dose group comparisons to Placebo p-value were based on the Wilcoxon-Mann-Whitney test. The Hodges-Lehmann nonparametric estimator was used to estimate the median difference between each PSL dose group versus placebo, along with the corresponding 95% CI of the estimate; Test type: Other; p = 0.316, Wilcoxon (Mann-Whitney) — Nominal p-values were not adjusted for multiplicity; Median Difference (Net) = 7.40, 95% CI 2-sided [-6.59 to 21.89]
Statistical Analysis 2: Comparison: Placebo (FAS) vs Padsevonil 100mg BID (FAS); [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.133, Wilcoxon (Mann-Whitney) — Nominal p-values were not adjusted for multiplicity; Median Difference (Net) = 9.99, 95% CI 2-sided [-3.15 to 23.26]
Statistical Analysis 3: Comparison: Placebo (FAS) vs Padsevonil 200mg BID (FAS); [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.203, Wilcoxon (Mann-Whitney) — Nominal p-values were not adjusted for multiplicity; Median Difference (Net) = 8.19, 95% CI 2-sided [-3.95 to 21.37]
Statistical Analysis 4: Comparison: Placebo (FAS) vs Padsevonil 400mg BID (FAS); [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.784, Wilcoxon (Mann-Whitney) — Nominal p-values were not adjusted for multiplicity; Median Difference (Net) = 2.39, 95% CI 2-sided [-13.65 to 17.79]

ADVERSE EVENTS:
Time Frame: Treatment-emergent AEs were collected from Baseline to Safety Follow-Up (up to Week 23)
Description: Adverse events refer to the SS which consisted of all participants who were administered at least 1 dose or a partial dose of IMP.
  TEAEs counts are for each study period: Treatment Period, Conversion Period for participants who entered the OLE study and Taper Period followed by SFU for participants not entering OLE study.
Groups:
- Placebo Treatment Period (SS): Participants randomized to the placebo group received 5-6 placebo tablets to maintain the blinding up to week 19. Participants formed the Safety Set (SS).
- Padsevonil 50mg BID Treatment Period (SS): Participants were randomized to receive a combination of tablets of padsevonil 50 mg and placebo (as appropriate) to maintain the blinding, bid up to week 19. Participants formed the SS.
- Padsevonil 100mg BID Treatment Period (SS): Participants were randomized to receive a combination of tablets of padsevonil 100 mg and placebo (as appropriate) to maintain the blinding, bid up to week 19. Participants formed the SS.
- Padsevonil 200mg BID Treatment Period (SS): Participants were randomized to receive a combination of tablets of padsevonil 200 mg and placebo (as appropriate) to maintain the blinding, bid up to week 19. Participants formed the SS.
- Padsevonil 400mg BID Treatment Period (SS): Participants were randomized to receive a combination of tablets of padsevonil 400 mg and placebo (as appropriate) to maintain the blinding, bid up to week 19. Participants formed the SS.
- Placebo Conversion Period (SS): A 3-week Conversion Period was required for study participants who chose to enroll in the open-label extension (OLE) study at the end of the 12-week Maintenance Period. Participants initially randomized to placebo progressively received padsevonil in a blinded way to reach the entry dose of 400mg/day for the OLE. Participants formed the Safety Set (SS).
- Padsevonil 50mg BID Conversion Period (SS): A 3-week Conversion Period was required for study participants who chose to enroll in the OLE study at the end of the 12-week Maintenance Period. The dose for participants initially randomized to padsevonil 50mg bid was gradually adapted (increased or decreased) in a blinded way to reach the entry dose of 400mg/day for the OLE. Participants formed the SS.
- Padsevonil 100mg BID Conversion Period (SS): A 3-week Conversion Period was required for study participants who chose to enroll in the OLE study at the end of the 12-week Maintenance Period. The dose for participants initially randomized to padsevonil 100mg bid was gradually adapted (increased or decreased) in a blinded way to reach the entry dose of 400mg/day for the OLE. Participants formed the SS.
- Padsevonil 200mg BID Conversion Period (SS): A 3-week Conversion Period was required for study participants who chose to enroll in the OLE study at the end of the 12-week Maintenance Period. The dose for participants initially randomized to padsevonil 200mg bid was gradually adapted (increased or decreased) in a blinded way to reach the entry dose of 400mg/day for the OLE. Participants formed the SS.
- Padsevonil 400mg BID Conversion Period (SS): A 3-week Conversion Period was required for study participants who chose to enroll in the OLE study at the end of the 12-week Maintenance Period. The dose for participants initially randomized to padsevonil 400mg bid was gradually adapted (increased or decreased) in a blinded way to reach the entry dose of 400mg/day for the OLE. Participants formed the SS.
- Placebo Taper and SFU Period (SS): A 4-week Taper Period was required for participants who chose not to enroll in the OLE study or who discontinued prior to the end of the 12-week Maintenance Period. Participants initially randomized to placebo group received 5-6 placebo tablets to maintain the blinding and have been gradually tapered off the IMP over a 3-week period followed by 1-week drug-free period.
  Afterwards, participants had a Safety Follow-Up visit 30 days after the last IMP intake. Participants formed the Safety Set (SS).
- Padsevonil 50mg BID Taper and SFU Period (SS): A 4-week Taper Period was required for participants who chose not to enroll in the OLE study or who discontinued prior to the end of the 12-week Maintenance Period. Participants initially randomized to padsevonil 50 mg bid have been gradually tapered off the IMP over a 3-week period followed by 1-week drug-free period. Afterwards, participants had a Safety Follow-Up visit 30 days after the last IMP intake. Participants formed the SS.
- Padsevonil 100mg BID Taper and SFU Period (SS): A 4-week Taper Period was required for participants who chose not to enroll in the OLE study or who discontinued prior to the end of the 12-week Maintenance Period. Participants initially randomized to padsevonil 100 mg bid have been gradually tapered off the IMP over a 3-week period followed by 1-week drug-free period. Afterwards, participants had a Safety Follow-Up visit 30 days after the last IMP intake. Participants formed the SS.
- Padsevonil 200mg BID Taper and SFU Period (SS): A 4-week Taper Period was required for participants who chose not to enroll in the OLE study or who discontinued prior to the end of the 12-week Maintenance Period. Participants initially randomized to padsevonil 200 mg bid have been gradually tapered off the IMP over a 3-week period followed by 1-week drug-free period. Afterwards, participants had a Safety Follow-Up visit 30 days after the last IMP intake. Participants formed the SS.
- Padsevonil 400mg BID Taper and SFU Period (SS): A 4-week Taper Period was required for participants who chose not to enroll in the OLE study or who discontinued prior to the end of the 12-week Maintenance Period. Participants initially randomized to padsevonil 400 mg bid have been gradually tapered off the IMP over a 3-week period followed by 1-week drug-free period. Afterwards, participants had a Safety Follow-Up visit 30 days after the last IMP intake. Participants formed the SS.
Arm/Group | Placebo Treatment Period (SS) | Padsevonil 50mg BID Treatment Period (SS) | Padsevonil 100mg BID Treatment Period (SS) | Padsevonil 200mg BID Treatment Period (SS) | Padsevonil 400mg BID Treatment Period (SS) | Placebo Conversion Period (SS) | Padsevonil 50mg BID Conversion Period (SS) | Padsevonil 100mg BID Conversion Period (SS) | Padsevonil 200mg BID Conversion Period (SS) | Padsevonil 400mg BID Conversion Period (SS) | Placebo Taper and SFU Period (SS) | Padsevonil 50mg BID Taper and SFU Period (SS) | Padsevonil 100mg BID Taper and SFU Period (SS) | Padsevonil 200mg BID Taper and SFU Period (SS) | Padsevonil 400mg BID Taper and SFU Period (SS)
All-Cause Mortality (participants affected / at risk) | 0/83 | 0/81 | 0/83 | 0/82 | 0/81 | 0/69 | 0/64 | 0/66 | 0/55 | 0/57 | 0/9 | 0/14 | 0/11 | 0/24 | 0/22
Serious Adverse Events (participants affected / at risk) | 3/83 | 5/81 | 4/83 | 3/82 | 5/81 | 0/69 | 0/64 | 0/66 | 2/55 | 0/57 | 1/9 | 1/14 | 0/11 | 0/24 | 0/22
Other Adverse Events (participants affected / at risk) | 45/83 | 54/81 | 60/83 | 53/82 | 65/81 | 11/69 | 18/64 | 10/66 | 5/55 | 5/57 | 3/9 | 3/14 | 0/11 | 3/24 | 4/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Treatment Period (SS) (N=83) | Padsevonil 50mg BID Treatment Period (SS) (N=81) | Padsevonil 100mg BID Treatment Period (SS) (N=83) | Padsevonil 200mg BID Treatment Period (SS) (N=82) | Padsevonil 400mg BID Treatment Period (SS) (N=81) | Placebo Conversion Period (SS) (N=69) | Padsevonil 50mg BID Conversion Period (SS) (N=64) | Padsevonil 100mg BID Conversion Period (SS) (N=66) | Padsevonil 200mg BID Conversion Period (SS) (N=55) | Padsevonil 400mg BID Conversion Period (SS) (N=57) | Placebo Taper and SFU Period (SS) (N=9) | Padsevonil 50mg BID Taper and SFU Period (SS) (N=14) | Padsevonil 100mg BID Taper and SFU Period (SS) (N=11) | Padsevonil 200mg BID Taper and SFU Period (SS) (N=24) | Padsevonil 400mg BID Taper and SFU Period (SS) (N=22)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Focal dyscognitive seizures (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure cluster (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Status epilepticus (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device battery replacement (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute psychosis (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Treatment Period (SS) (N=83) | Padsevonil 50mg BID Treatment Period (SS) (N=81) | Padsevonil 100mg BID Treatment Period (SS) (N=83) | Padsevonil 200mg BID Treatment Period (SS) (N=82) | Padsevonil 400mg BID Treatment Period (SS) (N=81) | Placebo Conversion Period (SS) (N=69) | Padsevonil 50mg BID Conversion Period (SS) (N=64) | Padsevonil 100mg BID Conversion Period (SS) (N=66) | Padsevonil 200mg BID Conversion Period (SS) (N=55) | Padsevonil 400mg BID Conversion Period (SS) (N=57) | Placebo Taper and SFU Period (SS) (N=9) | Padsevonil 50mg BID Taper and SFU Period (SS) (N=14) | Padsevonil 100mg BID Taper and SFU Period (SS) (N=11) | Padsevonil 200mg BID Taper and SFU Period (SS) (N=24) | Padsevonil 400mg BID Taper and SFU Period (SS) (N=22)
Vertigo (Ear and labyrinth disorders) | 7 (7) | 3 (3) | 2 (2) | 3 (3) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (7) | 4 (4) | 7 (7) | 2 (3) | 7 (13) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 6 (8) | 3 (4) | 5 (7) | 4 (5) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 10 (10) | 20 (27) | 12 (17) | 14 (22) | 20 (21) | 3 (3) | 5 (5) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (5) | 5 (5) | 9 (13) | 7 (11) | 5 (5) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (3) | 5 (5) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 4 (4) | 2 (2) | 1 (1) | 1 (2) | 7 (7) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anticonvulsant drug level increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 9 (9) | 18 (19) | 23 (31) | 19 (25) | 28 (55) | 3 (3) | 2 (2) | 1 (1) | 2 (2) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 10 (11) | 19 (24) | 24 (29) | 25 (26) | 30 (35) | 1 (1) | 4 (5) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 10 (14) | 17 (29) | 9 (16) | 15 (21) | 9 (31) | 0 (0) | 3 (3) | 2 (3) | 0 (0) | 1 (5) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1) | 8 (9) | 14 (14) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 5 (5) | 2 (2) | 6 (6) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 1 (2) | 3 (3) | 3 (3) | 5 (5) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nystagmus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 8 (8) | 4 (4) | 7 (7) | 1 (1) | 5 (6) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3) | 1 (1) | 1 (2) | 7 (9) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paranoia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-10-12): https://cdn.clinicaltrials.gov/large-docs/83/NCT03373383/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-12): https://cdn.clinicaltrials.gov/large-docs/83/NCT03373383/SAP_001.pdf